CLINICAL TRIAL: NCT03966287
Title: Analysis of Pain and Quality of Life in Patients With Charcot-Marie-Tooth Neuropathy (CMT)
Status: Completed | Type: Observational
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Michael W Sereda, MD, Professor of Neurology, Prof. Dr. Michael W. Sereda, University Medical Center Goettingen
Other Study IDs: 02202
Record Dates: First submitted 2019-05-21; First posted 2019-05-29 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: CMT

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to qualitatively and quantitively evaluate pain in patients suffering from CMT with 3 standardized questionnaires (SF-36, NPSI-G, PAIN DETECT) as well as its impact on the quality of life.

DETAILED DESCRIPTION:
Hereditary neuropathies are a group of clinically and genetically heterogeneous diseases of the peripheral nervous system. Charcot-Marie-Tooth disease (CMT), also known as hereditary motor and sensory neuropathy (HMSN), is the most common form of hereditary neuropathy with a prevalence of approximately 1 in 2,500 and with approximately 30,000 affected persons in Germany. There is no therapy known so far. In addition to the characteristic symptoms of a distal to proximal progressive symmetric muscular atrophy, especially of the lower extremities, there is a weakening of the muscles of the lower legs and feet, with emphasis on the "small" foot muscles and the peroneal muscle group, which clinically manifests as a so-called "stepper gait". It is also known that many CMT patients additionally suffer from pain, but more detailed studies on pain quality and quantity and their impact on patients' quality of life have not yet been systematically performed. These parameters will be investigated in this study, supported by the company Grünenthal, in the form of a questionnaire survey with validated questionnaires on pain and quality of life for at least 200 CMT patients. A representative result could lead to further investigations of pain in CMT patients and ultimately to the development of an adequate pain therapy.

Recruitment of patients will occur mainly through a call of the Germany-wide CMT registry, which is part of the national research network CMT-NET (coordinator: Prof. Michael Sereda). Interested patients are invited to contact the study team at the UMG. The patients will be informed about the study and if further interested 4 questionnaires (1 regarding the personal history as well as 3 standardized questionnaires from literature regarding quality of life and pain (SF-36, NPSI-G, PAIN DETECT) will be sent to the patients together with obligatory study documents and a pre-franked return envelope. A personal visit at the UMG is not planned, so that the patients don´t have any expenses. The data are pseudonymized at the UMG and transferred to a database and finally statistically evaluated by Gruenenthal.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of CMT
* Genetic confirmation of CMT diagnosis
* Age between 18 and 65 years
* Signed consent form

Exclusion Criteria:

* Other relevant neurological or psychiatric diseases, acute or past
* Serious internal medical illness
* Drug and / or alcohol dependence
* Participation in another clinical trial within 4 weeks prior to enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: German-wide, registered patients in CMT-registry
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
SF-36 Questionnaire | 1 year
  Questionnaire to evaluate health status
NPSI-G Questionnaire | 1 day
  Questionnaire to discriminate neuropathic and non-neuropathic pain
PAIN DETECT Questionnaire | 4 weeks
  Questionnaire for the diagnosis of neuropathic pain (intensity, pattern, quality)

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre, Goettigen, Germany